CLINICAL TRIAL: NCT03184441
Title: Premie Pouch to Manage Deformational Plagiocephaly in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Boston Orthotics & Prosthetics (Other)
Responsible Party: Principal Investigator, Michele DeGrazia, Director of Nursing Research, Neonatal Intensive Care Unit, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00011098
Record Dates: First submitted 2017-04-28; First posted 2017-06-12 (Actual); Results first posted 2018-08-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-07

CONDITIONS: Plagiocephaly
MeSH Terms: conditions — Plagiocephaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Premie Pouch (Experimental): All participants will receive the experimental treatment with the Premie Pouch device.
  Interventions: Device: Premie Pouch

INTERVENTIONS:
Device: Premie Pouch — The Premie Pouch is an experimental device meant to manage the development of Deformational Plagiocephaly (DP) starting immediately following birth. The Premie Pouch has a concave-shaped foam insert that will provide a resting surface for the infant's head and body that will eliminate uneven pressure on the infant's occiput while maintaining correct body alignment. Also, the posterior neck area of the infant will be supported by a fixed bridge section of the foam insert. The Premie Pouch is designed specifically for the very low birth weight (VLBW) infant.

SUMMARY:
This pilot project proposes to develop and test a new device to manage (defined as resolving, prohibiting, inhibiting or preventing) the development of Deformational Plagiocephaly (DP) in prematurely born infants weighing < 1 kilogram.

DETAILED DESCRIPTION:
Prematurely born infants are prone to developing Deformational Plagiocephaly (DP), a flattened head shape from repeatedly being positioned in the same direction while on a flat or solid surface. Left untreated approximately 30-40% of infants retain this abnormal head shape at 3-4 years of age. According to reports DP has the potential to affect the infant's social and neurobehavioral development.

Recent research on the PlagioCradle™ device demonstrates prevention and correction of DP in hospitalized infants. However, extremely premature infants, weighing < 1 kilogram cannot use the device known as the PlagioCradle™. This device only accommodates infants weighing > 1 kilogram. When infants eventually reach 1 kilogram, healthcare providers have trouble fitting them to the smallest version of the PlagioCradle™ device and must place the infant in a layer meant for a larger infant. Use of the larger layer often requires that infants' lay in a side-lying position until their head shapes begin to improve. It is more desirable that infants be placed in the appropriate layer so that they may be positioned supine, prone, side-lying left and right, to ensure optimal development. This pilot project proposes to develop and test a new device to manage (defined as resolving, prohibiting, inhibiting or preventing) the development of DP in prematurely born infants weighing < 1 kilogram.

NICU (Neonatal Intensive Care Unit) nurses have used waterbed therapy, air-filled mattresses, foam mattresses and repositioning procedures in an attempt to manage the development of DP, but these methods have had limited success. The reason these devices are not successful is because they do not provide structure or support for the soft cranium that has un-fused sutures and that have not become fixed or solidified. As a result, the soft, malleable cranium then takes the shape of the bedding or device it is placed upon, which is usually flat (including the aforementioned positioning devices).

The PlagioCradle™ (previously known as the cranial cup) is an orthotic device developed by Gary Rogers M.D., J.D., M.B.A., M.P.H., a craniofacial surgeon formerly of Boston Children's Hospital and James Miller C.P.O. a licensed orthotist. The PlagioCradle™ is an anatomically correcting, repeatedly adjustable, concave-shaped resting surface for an infant's head and body that effectively eliminates uneven pressure on the infant's occiput while maintaining correct body alignment. In addition, the posterior neck area of the infant is supported by a fixed bridge section, which also serves to off-load or reduce contact pressure between the rest surface and the occiput, especially as the cavity of the device deepens. The PlagioCradle™ has been found to be an effective tool in preventing or correcting DP in preterm and term infants. The PlagioCradle™ accommodates infants weighing 1 Kg or larger.

The Premie Pouch is meant to serve as precursor to the PlagioCradle™ by managing the development of DP starting immediately following birth. Like the PlagioCradle™, the concave-shaped foam insert will provide a resting surface for the infant's head and body that eliminate uneven pressure on the infant's occiput while maintaining correct body alignment. Also, the posterior neck area of the infant will be supported by a fixed bridge section of the foam insert. However the Premie Pouch is designed specifically for the VLBW infant.

The rectangular shaped Premie Pouch device measures approximately 10X15 inches in size. The cover is made of a stretchy, washable fabric such as jersey or fleece. There are two pockets; one to accommodate a foam insert and another will accommodate a bladder insert of soft squishy pellets. The Premie Pouch will come with two cotton/Velcro positioning straps that can be used to provide containment of the infant's arms and/or legs, adding to their comfort when using the device.

Pocket #1 will accommodate a foam insert. Nurses will select one of 3 different sized pre-molded foam inserts, sized for infants weighing < 1 Kg. Once the appropriate insert is selected it will be placed inside pocket #1. As the infant's grows, nurses can select a new insert so that a neutral position is maintained and the head sits comfortably in the depression. When appropriately sized the head can move freely and a small gap, approximately 1/8th inch, will be noted around the head.

The foam insert will facilitate a normalized head shape by providing structure to the cranium. Border stitching of the cover around the foam will keep the insert in place when the device is moved. Infants can be positioned supine or side lying when using the top layer of the device holding the foam insert. The bottom layer of the device will be used for prone positioning when the foam insert is removed Pocket #2, the bottom layer of the Premie Pouch will contain a bladder of soft squishy pellets that offer a comfortable place for infants to rest when positioned prone (but that also remains in place when using the top layer with the insert in place). To use this layer of the device, the nurse need only remove the foam insert.

The Premie Pouches are to be constructed by an experienced seamstress hired to sew the devices and the bladder inserts that contain the pellets. Three foam inserts (each with a slightly different depression depth to ensure a semi customized fit) will be provided for use with each Premie Pouch device, along with three cotton covers Premie Pouch Care and Maintenance. Each infant participant will receive a new device and 2 extra sets of covers. The outer covering of the device can be laundered either by a laundry service or the infant's mother. The foam inserts and bladder inserts (housed in a water repellent polymer-coated fabric) will be able to be wiped down using antibacterial wipes routinely used for cleaning similar devices in the participating NICUs. The covers of the device are made of cotton/spandex blend.

Purpose and Specific Aims:

Technological improvements such as advanced MRI techniques allow researchers to detect diminutive changes in brain structure on infants with positional head shape deformities. In addition new developmental assessments allow researchers to detect a spectrum of neurobehavioral and motor development problems. These type of advances have allowed researchers to establish a relationships between DP, neurobehavioral problems and auditory processing disorders. These relationships suggest that DP may be more problematic than once thought, hence the need for preventative measures.

At present time, nurses in NICU's across the nation manage DP by repositioning their patient's, as frequently as their condition permits, and with the use of gel pillows and other positioning aids like the Z flo. In this study the investigator is taking a proactive approach toward DP management through development of the Premie Pouch and investigation of its safety, feasibility and very preliminary information on its effectiveness.

Research questions:

Question 1. Is the Premie Pouch safe for use with premature infants weighing < 1 Kg as evidenced by the absence of adverse events? Question 2. Is the Premie Pouch feasible for use with premature infants weighing < 1 Kg as measured by the number of hours of use per day on the device? Question 3. Do bedside nurses caring for the study infant's rate the Premie Pouch easy to use? Question 4. What is the relationship between time (as measured in hours) spent on the Premie Pouch with the foam layer in place and head shapes (as measured by cranial index and cranial symmetry) in a sample of premature infants weighing < 1 Kg?

Education:

Research Staff- Prior to the initiation of study procedures all research personnel will be Citi program trained. Also all study staff will receive training by the researcher or key study personnel on all study procedures and the use of the positioning device. During training, emphasis will be placed on procedures to ensure the safe use of the positioning device and procedures to ensure patient safety during head shape measures. A Manual of Operations at each study site will include directives for obtaining the head shape measures and examples of appropriate documentation on the data collection tools.

NICU Staff- Prior to enrollment of study subjects or the initiation of any study procedures, staff in the NICUs will receive education on the use of the Premie Pouch device and on their role during the study. The NICU staff will also be given the opportunity to have any questions answered. A Manual of Operations will be provided to each of the NICUs that will store copies of the study protocol, consent, procedure for obtaining head shape measures and instructions on use, care and maintenance of the study device.

Parent- Study staff will be responsible for educating parents about the study and reeducating them as needed during the course of their infant's participation.

Enrollment: Once the infant is in a critical but stable condition (which usually happens in the first two weeks of life), a member of the medical or nursing staff will ask the parent(s) of prospective study subjects if they are interested in hearing about this research study. If the parent(s) agree the researcher or study staff member trained in obtaining consents will approach them to explain the study. In addition, the researcher or study staff member will provide the parent(s) with written materials that describe the study and their infant's involvement. The parent(s) will be given the opportunity to ask questions. If the parent(s) agree to participate they will be asked to sign an informed consent and HIPPA form.

Procedures:

All participants will receive the experimental treatment with the Premie Pouch. While using the device, nurses will (as per unit routines) routinely reposition infants every 3 to 4 hours minimum, including prone. Nurses will utilize the Premie Pouch device whenever the infant is on the warmer, in the isolette or bed, unless specific procedures or medical interventions preclude it use. Nurses will be instructed to reposition infants frequently, ensuring that infants spend (equal time) approximately 1/2 of the day supine (or side lying) on the foam layer of the device. Nurses will be instructed to document device use on the daily positioning logs for the length of the study. Study staff will monitor device use, ensuring that the daily positioning logs are being completed.

Repositioning infants every 3-4 hours minimum, is an important aspect of neonatal care. In addition to facilitating a normal head shape, repositioning helps to facilitate good skin integrity, skeletal development, biomechanical alignment, and provides exposure to proprioceptive, tactile, and visual stimuli. Similar to other positioning devices used in this population, long velcro straps (rough side up) that wrap around the device and the infant, will provided with the Premie Pouch device. Nurses can apply these straps to gently secure arms and legs in a comfortable position.

Once the infant participants reach 1 Kg and outgrow the Premie Pouch device, participation in this study will end. At that time nurses will care for the infants using routine positioning techniques and devices available in the respective unit (such as but not limited to gel pillows and other positioning aids like the Z flo or Plagiocradle.

ELIGIBILITY:
Inclusion Criteria:

1. Infants weighing </= 900 grams. (Selecting a weight below the 1 Kg cut off for using the device will allow the infant an opportunity to use the device before outgrowing it.)
2. Infants born at >/= 22 weeks gestation.
3. Infants </= 40 days of age at enrollment.
4. Infants that receive medical clearance from their healthcare team.
5. Infants that have an estimated minimum hospital length of stay = / > 14 days from the time of enrollment.
6. Every effort will be made to include infants from non-English speaking families as long as using all available resources; the parents can successfully communicate with the research team. The research team will utilize interpreter services and other resources (immediate family members and supports) to facilitate this process when applicable.

Exclusion Criteria:

1. Infants that require only prone positioning to maintain airway patency (such as those with Pierre Robin Syndrome/Sequence) will not be eligible to participate; this is because infants must be able to lie supine for at least part of the day.
2. Infants requiring medical devices such as a continuous ventricular drain, subgaleal shunt, or intravenous catheters (unless placement of the IV is temporary) as they prevent proper positioning using the Premie Pouch.
3. Infants with a craniofacial anomaly, craniosynostosis, cervical anomaly, or critical airway.
4. Infants with Cutis Aplasia or significant skin breakdown to the scalp, because the experimental device may worsen a preexisting condition.
5. Infants that are to be transferred to a non-participating hospital within 14 days of enrollment as this timeframe may not allow adequate evaluation of the Premie Pouch.

Max Age: 40 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele DeGrazia, PhD, NNP, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seruya M, Oh AK, Sauerhammer TM, Taylor JH, Rogers GF. Correction of deformational plagiocephaly in early infancy using the plagio cradle orthotic. J Craniofac Surg. 2013 Mar;24(2):376-9. doi: 10.1097/SCS.0b013e31828010d1. PMID 23524697
- [Background] Rogers GF, Miller J, Mulliken JB. Comparison of a modifiable cranial cup versus repositioning and cervical stretching for the early correction of deformational posterior plagiocephaly. Plast Reconstr Surg. 2008 Mar;121(3):941-947. doi: 10.1097/01.prs.0000299938.00229.3e. PMID 18317143
- [Background] DeGrazia M, Giambanco D, Hamn G, Ditzel A, Tucker L, Gauvreau K. Prevention of deformational plagiocephaly in hospitalized infants using a new orthotic device. J Obstet Gynecol Neonatal Nurs. 2015 Jan-Feb;44(1):28-41. doi: 10.1111/1552-6909.12523. Epub 2015 Jan 8. PMID 25573141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 3 study sites (i.e. Neonatal Intensive Care Units). 6/30/16-7/30/16.
Groups:
- Premie Pouch: All participants will received the experimental treatment with the Premie Pouch device.
  Premie Pouch: The Premie Pouch is an experimental device meant to manage the development of Deformational Plagiocephaly (DP) starting immediately following birth. The Premie Pouch has a concave-shaped foam insert that will provide a resting surface for the infant's head and body that will eliminate uneven pressure on the infant's occiput while maintaining correct body alignment. Also, the posterior neck area of the infant will be supported by a fixed bridge section of the foam insert. The Premie Pouch is designed specifically for the very low birth weight (VLBW) infant.
Period: Overall Study
Arm/Group | Premie Pouch
Started | 11
Completed | 10 (Last subject completed study)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Premie Pouch
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: days] | 17.9 [5 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Cranial Abnormalities Were Measured at Enrollment [Number; unit: participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety of Use of the Premie Pouch in VLBW Infants
Description: Frequency of participants with adverse events reported using the Premie Pouch Adverse Event Data Collection Tool.
Time Frame: From date of enrollment to date of study completion (range 19-47 days)
Population: Participants with adverse events
Measure: Number; unit: participants
Groups:
- All Subjects Recieved the Study Device: Clinical decompensation of one subject, not device related, and not included in analysis. Did not meet minimal data requirement.
Arm/Group | All Subjects Recieved the Study Device
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Feasibility of Use of the Premie Pouch in VLBW Infants
Description: Documented hours per day (24 hours) on the Premie Pouch device
Time Frame: Number of hours per each 24 hour period on the device
Population: Hours on device per day
Measure: Mean (Full Range); unit: hours per day
Arm/Group | Premie Pouch
Number analyzed (Participants) | 10
hours per day | 20.1 [14.2 to 23.3]

3. Secondary Outcome: Number of Participants With Normal Cranial Index
Description: Cranial index (An objective front to back and side to side, measure that quantifies head shape by dividing head width by length then multiplying it by 100%) for each of participants was measured at study completion. Participants falling within the normal range of 73%-85% had normal cranial index.
Time Frame: Cranial index at study completion
Population: Normal cranial index at study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Premie Pouch
Number analyzed (Participants) | 10
Participants | 5

4. Secondary Outcome: Number of Participants With Normal Cranial Symmetry
Description: To assess for cranial asymmetry of the head shape at study completion, the right anterior-posterior measures and left anterior-posterior measures of infant's head shapes were obtained. Cranial symmetry was defined as less than 8mm difference in the right and left anterior-posterior measures.
Time Frame: Cranial symmetry at study completion
Population: Normal Cranial Symmetry
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Recieved the Study Device: All participants will received the experimental treatment with the Premie Pouch device.
  Premie Pouch: The Premie Pouch is an experimental device meant to manage the development of Deformational Plagiocephaly (DP) starting immediately following birth. The Premie Pouch has a concave-shaped foam insert that will provide a resting surface for the infant's head and body that will eliminate uneven pressure on the infant's occiput while maintaining correct body alignment. Also, the posterior neck area of the infant will be supported by a fixed bridge section of the foam insert. The Premie Pouch is designed specifically for the very low birth weight (VLBW) infant.
Arm/Group | All Subjects Recieved the Study Device
Number analyzed (Participants) | 10
Participants | 10

5. Secondary Outcome: Premie Pouch Ease of Use
Description: This the percentage or nurses that found the Premie Pouch device easy to use.
Time Frame: From date of enrollment to date of study completion (range 19-47 days)
Measure: Count of Participants; unit: Participants
Groups:
- Premie Pouch: Nurses caring for participants in the study
Arm/Group | Premie Pouch
Number analyzed (Participants) | 23
Participants | 18

ADVERSE EVENTS:
Arm/Group | Premie Pouch
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No